CLINICAL TRIAL: NCT01434264
Title: Cross-disciplinary Evaluation of Efficacy and Effectiveness of Individualized Complementary Therapies: Evaluating Personalized Effect of Energy Healing as an Individualized Intervention
Brief Title: Evaluating Personalized Effect of an Individualized Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Aarhus (Other); The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Principal Investigator, Helle Johannessen, Professor, mag.scient., PhD, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-065176/DSF
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Cancer
Keywords: rehabilitation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Spiritual Therapies; Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Self-selected energy healing (Experimental): Self-selected healing in the self-selection arm
  Interventions: Procedure: Energy healing
- self-selected control (No Intervention): Self-selected control in the self-selection arm
- randomized to energy healing (Experimental): Randomized to healing in the randomization arm
  Interventions: Procedure: Energy healing
- Randomized control (No Intervention): Randomized to control in the randomization arm

INTERVENTIONS:
Procedure: Energy healing — "Healer-Ringen", a Danish national association of healers, selects healers with an educational background as required by the Registry of Alternative Practitioners (RAB) and have rooms reserved for the healing practice. The treatment takes place in the clinic of the healer and is not restricted in respect to what form of energy healing that shall be used, provided that it is based on the idea of the healer providing some kind of energy by the hands to the participant. Conversation as usual is accepted, but no other form of therapy may be provided. The intervention consists of four sessions over a period of two months, distributed as decided by each participant-healer pair.
  Other Names: Spiritual healing; Reiki
  Arms: Self-selected energy healing; randomized to energy healing

SUMMARY:
Energy healing is among the most commonly used forms of complementary and alternative medicine among cancer patients. There are, however, few studies on the effects of energy healing for cancer and cancer associated symptoms and none of them are of a volume or quality that allows reliable conclusions to be drawn. Qualitative studies on energy healing in Denmark have demonstrated that the interventions are individualized and the expected outcomes personalized. This research points to the need for a research design that can evaluate personalized outcomes of individualized treatments and at the same time adhere to general demands of external and internal validity.

The objective of this study is to test the effectiveness of energy healing as an individualized rehabilitative intervention to improve outcomes of personal choice among persons who have completed a conventional intended curative treatment for colorectal, breast and prostate cancer. The study is designed as a pragmatic clinical trial with personalized outcomes.

The study attempts to maximize external validity by using a design that incorporates important features of energy healing administered in real-life settings: 1a) allowing participants self-selection to healing and non-healing control, 1b) assessing individual participant-selected treatment goals, 1c) allowing the treatment to be performed in the private clinics of the healers. To maximize internal validity similar to that obtained in a randomized, clinical trial design, the study will 2a) randomize participants to self-selection and randomized groups of intervention and control; and 2b) supplement the assessment of personalized treatment goals with assessment of outcomes with standardized measures.

The study will account for a number of possible moderators of the effects, including 3a) socio-demographics and 3b) previous experience with complementary and alternative treatment. Outcome measures will be assessed by questionnaires, physical measurements, data from administrative registries as well as semi-structured interviews and participant observation. Possible patterns in the various forms of data will be examined for concordances and discrepancies.

Finally, the methods will be discussed in terms of their generalizability as a model for evaluating personal outcomes of individualized treatments with high levels of external and internal validity.

DETAILED DESCRIPTION:
PRIMARY OUTCOMES AND HYPOTHESES

The primary outcome is to investigate whether "energy healing" as an individualized form of treatment can improve personal concerns identified by the individual patient in the MYCaW questionnaire.

Hypotheses:

* The effects found will be larger for the primary, personalized, outcomes (MYCaW) than when assessed with standardized measures.
* Patients that self-select energy healing will experience larger effects for primary outcomes than patients that randomized to the intervention.
* The primary, personalized outcomes will change more during the course of the treatment in the intervention groups than in the control groups.

SECONDARY OUTCOMES AND HYPOTHESES

Secondary outcomes concern three independent but related areas: (1) Will energy healing have a statistically significant (p < 0.05) effect on secondary outcomes assessed with standardized, validated instruments, including physical health survey, physical activity, cancer-related QoL, depressive symptoms, and mood? (2) Will energy healing have a positive impact on daily physical performance as subjectively described in dairies? (3) Will energy healing influence participants' subjective experience of their illness and recovery? (4) Will energy healing influence participants' self-reported burden of late effect after cancer treatment?

Hypotheses:

* No significant effects of healing on secondary, standardized, outcomes (Physical health survey, physical activity, QoL, Depressive symptoms, mood) are anticipated.
* No significant effect on levels of daily physical performance as reported in diaries is anticipated.
* Participants that self-select energy healing will report significantly larger effects on secondary outcomes than patients randomized to intervention.
* No significant effect on participants' self-reported burden of late effects is anticipated.

Further, it is expected that the qualitative analysis will inform whether the energy healing provides participants with images that are embodied in their perception of self, illness and recovery and whether this is acknowledged by participants as meaningful for them in the particular situation in which they are embedded.

HYPOTEHSES RELATED TO MEDIATION AND MODERATION OF EFFECTS

A number of factors are anticipated to mediate and moderate the effects of energy healing.

Hypotheses:

* The effect of healing will be larger, if participants o report higher levels of "absorption" (i.e. "openness to experience")

  * report higher expectations of benefits
  * report previous positive experience with CAM
  * report a positive attitude towards CAM
  * report prior experience with energy healing
  * report faith in God or a higher spiritual power
  * experience a better healer-patient relationship
* Those that change their primary selected outcome over the course of treatment will score higher on the questionnaire relating to the healer-patient relationship.

Further, it is expected that the qualitative analysis will shed light on whether and how

* participants subjectively express a change in their perception of self and illness corresponding with the healer's recommendations;
* ritualization of the healing session provides for participants' subjective acknowledgement of the healer-patient relationship;

The quantitative and qualitative data in combination are expected to confirm the following hypothesis:

* If the healer is able to ritualize, orchestrate and 'key' the performance of the healing ritual by means of stylistic devices as e.g. the burning of incense, music, etc., and if he/she is a skilled symbol manager, and if the participant subjectively acknowledge these aspects, the participant will score high on standardized questionnaires.

TERTIARY OUTCOMES

Finally, a number of issues will be explored relating to the value attributed to the treatment by the participants. It will be explored:

* How much money are the participants in the intervention groups willing to spend on this kind of therapy
* How far a distance participants are willing to drive to receive this kind of therapy

STUDY DESIGN

The study is a pragmatic trial allowing healers to adjust the intervention (energy healing) to each participant and to undertake treatment-related communication as usual. The study is designed to allow for analysis of the implications of self-selection by randomizing participants to a self-selection arm and a randomized arm, each arm with corresponding control groups. Finally, the study design allows participants to identify what they consider to be their primary outcomes by using open outcome forms and semi-structured interviews in conjunction with validated, standard measures. In order to encompass the expected variation in primary outcomes and to investigate the interrelations of different types of outcomes, the study is designed as a cross-disciplinary investigation.

RECRUITMENT

125 persons for the treatment groups and 200 persons for the control groups will be recruited in two ways; 1) Lists of patients who have completed their hospital treatment for colorectal, breast and prostate cancer within the last 12 months will be extracted from The National Patient Registry, and, 2) lists of patients who have completed intended curative treatment for colorectal cancer within the last month will be provided by the involved hospital departments from the Region of Southern Denmark. All patients considered eligible are randomized to self-selection arm (SSA) or randomization arm (RA) and mailed: 1) A letter inviting them to participate in the study, 2) Information about the study and the group they are assigned to, 3) A baseline questionnaire, 4) An informed consent form, allowing them to be contacted by the research team and a healer, and 5) A pre-paid return envelope. All invited persons are then contacted by telephone in order to answer any questions they may have concerning the study. Persons willing to participate are asked to complete the baseline questionnaire and the informed consent form and return these. Persons who are unwilling to participate will be asked for the reasons and a drop-out register will be established. After two consecutive reminder calls and no response, a participant will be considered a drop-out (see Figure 1).

After allocation of participants to healers, the healers are contacted by telephone and letter with information on the participants and repetition of the procedure to be followed. The healers will arrange contacts to the participants who have been assigned to receive energy healing within two days in order to agree on a date for the first session.

All project procedures will be administered and organized using an encrypted ACCESS database aligned with the study protocol procedures. Day-to-day data collection activities will thus be based on computerized enquiries, and all procedural and unplanned events, such as i.e. patient telephone calls, will be registered.

RANDOMIZATION

Possible participants are initially and before the first contacts randomized to SSA and RA by a centralized, computerized procedure, e.g. the Minim (Minimisation Program for Allocating Patients to Treatments in Clinical Trials). Stratified; The sample will be stratified according to type of cancer and gender.

Following the reception of baseline questionnaires and informed consent form from the group randomized to the RA, the RA is further randomized to intervention and control groups by a similar procedure.

ASSESSMENT

Questionnaires:

Baseline questionnaires will be administrated before first treatment. Additional questionnaire packages will be administered to the participants 10 days, 10 weeks and 18 weeks after baseline. Additionally, those in the healing intervention groups complete questionnaire packages immediately before and after their third healing session. For comparison the control groups complete a questionnaire package 6 weeks after baseline.

Diaries:

20 participants from each of the four groups are asked to fill in an activity diary (conc. activities from sleep to strenuous activity) and time consumption (minutes and hours) during the day. The activity diary will be completed for seven days at baseline, seven days at week 10 and seven days at week 18.

Qualitative semi-structured interviews:

8 participants from each of the two intervention groups and control groups will be included for qualitative interviews and participant observation. The interviews and participant-observation will be conducted before and after the treatments and enable comparison of dispositions and processes of change. Interviewees will be selected to ascertain distribution in age and previous use of CAM (particularly energy healing). All interviews will be recorded if the participants are comfortable with it.

Participant-observation:

12 participants will be followed with 1 day's participant-observation before the first treatment and 2 days' participant-observation after the final treatment in settings, which the patient consider as important domains in his/her life and in the 'returning-to-life' process. Further, participant-observation will be conducted in some of the clinics involved in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of colorectal, breast and prostate cancer
2. Completed treatment with intended cure and no current cancer

Exclusion Criteria:

1. Unwillingness to comply with data collection protocol
2. Mentally and cognitively incapable to participate in the study
3. Poor understanding and expression of the Danish language
4. In palliative care or cancer recurrence prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in personal concerns identified by the patient in the MYCaW questionnaire. | Measured 10 days after baseline, 6 weeks after baseline (before third treatment), 10 weeks and 18 weeks after baseline
  The primary outcome is to investigate whether "energy healing" as an individualized form of treatment can improve personal concerns identified by the patient in the MYCaW questionnaire.

SECONDARY OUTCOMES:
Changes in Physical Health Survey | 10 days, 10 weeks and 18 weeks after baseline
  Late complications
Changes in SF-36 Physical activity | 10 days, 10 weeks and 18 weeks after baseline
  Physical activity
Changes in Facit-sp QoL | Baseline, 10 weeks and 18 weeks after baseline
  Physical, emotional, social and spiritual well-being
Changes in BDI-II depressive symptoms | Baseline, 10 weeks and 18 weeks after baseline
  Depressive symptoms
Changes in POMS Mood | Baseline, 6 weeks after baseline (before and after third treatment), 10 weeks and 18 weeks after baseline
  Profile of mood states
Changes in Daily physical performance | 10 days, 10 weeks and 18 weeks after baseline
  Daily physical performance as reported in diaries

CONTACTS AND LOCATIONS:
Overall Officials: Helle Johannessen, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Christina Gundgaard Pedersen, Aarhus, Denmark

REFERENCES:
- [Derived] Agdal R. "Is the Pain a Sign of Healing?": Cancer Patients' Experiences of Energy Healing in a Pragmatic Trial. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221118328. doi: 10.1177/15347354221118328. PMID 36154510